CLINICAL TRIAL: NCT07061197
Title: Effect of Communicating Structured Benefit and Harm Information in European Patient Leaflets on Individuals' Expectations About New Medicines: a Randomized Controlled Trial
Brief Title: Effect of Communicating Structured Benefit and Harm Information in European Patient Leaflets on Individuals' Expectations About Medicines
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Economics and Political Science (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 494342
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Cancer
Keywords: Cancer; Prescription drug information
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (standard patient leaflet) (Placebo Comparator)
  Interventions: Other: Control (standard patient leaflet)
- Patient leaflet with the EMA's proposed key information section including qualitative statements (Experimental)
  Interventions: Other: Patient leaflet with the EMA's proposed key information section including qualitative statements.
- Patient leaflet with a key information section providing qualitative and quantitative information (Experimental)
  Interventions: Other: Patient leaflet with a key information section providing both qualitative and quantitative information on drug benefits and harms.

INTERVENTIONS:
Other: Patient leaflet with the EMA's proposed key information section including qualitative statements. — The standard patient leaflet supplemented with a key information section. This section included qualitative descriptions of the goal of treatment, the main benefits, contraindications, and the most serious side effects. The content was designed to reflect the EMA's proposed format for improving the patient information leaflet.
  Arms: Patient leaflet with the EMA's proposed key information section including qualitative statements
Other: Control (standard patient leaflet) — The standard patient information leaflet for a recently approved cancer drug, tivozanib (Fotivda), obtained electronically from the EMA website. The standard patient information does not contain structured benefit information.
  Arms: Control (standard patient leaflet)
Other: Patient leaflet with a key information section providing both qualitative and quantitative information on drug benefits and harms. — The standard patient leaflet, supplemented with a key information section including quantitative data on the drug's main benefits and side effects, presented in a summary table format. This section provided structured information about the indication and goal of treatment, how the drug was studied (the comparator treatment and number of patients enrolled in the clinical trial that supported the drug's approval), and data on the drug's benefits and side effects.
  Arms: Patient leaflet with a key information section providing qualitative and quantitative information

SUMMARY:
This online randomized controlled trial will evaluate whether adding a key information section to patient information leaflets leads to more accurate expectations and improves participants' understanding. We will test the impact of including quantitative information on drug benefits in addition to qualitative statements, versus including qualitative statements only. Participants will be randomly assigned to one of three groups: (1) a standard patient leaflet that contains no information on drug benefits, (2) a leaflet featuring a key information section that includes qualitative statements about drug benefits, or (3) a leaflet featuring a key information section that includes quantitative information about drug benefits in addition to qualitative statements.

DETAILED DESCRIPTION:
Currently, European legislation requires that patient information leaflets accompanying all prescription medicines list the adverse effects of the medicine and provide guidance on its safe and appropriate use. In 2025, the European Medicines Agency (EMA) launched a public consultation on a proposal to include a new 'key information section' in the patient leaflets across Europe. A key information section is intended to help users quickly access non-promotional information about both the drug benefits and risks of a drug.

This study aims to evaluate the effect of including information about drug benefits, either qualitatively or both qualitatively and quantitatively, on individuals' expectations of a new cancer drug, using the European patient leaflet.

In this online randomized controlled trial, a nationally representative sample of adults from the United Kingdom will be randomly assigned to 1 of 3 versions of a patient leaflet: (1) the standard patient information leaflet (control), (2) a leaflet with the EMA's proposed key information section containing qualitative statements, or (3) a leaflet with a key information section providing both qualitative and quantitative data on the drug's benefits and harms. The patient leaflet used in the study was for a cancer drug (tivozanib).

The primary outcome is participants' expectations regarding the drug's benefits and harms. Secondary outcomes include participants' understanding of the information, participants perceived magnitude of the drug's benefits and harms, and their satisfaction with the leaflet content.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age and older,
* Adults fluent in English,
* Adults residing in the United Kingdom (i.e., nationally representative sample of UK adults).

Exclusion critera:

- Participants who do not meet all 3 inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2100 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Expectations | Assessed during 15-minute survey.
  Multiple choice questions assessing expectations about the benefits of tivozanib, a cancer drug approved by the European Medicines Agency.
  For example, "does Fotivda cure advanced kidney cancer?" Measured on a 4 point-Likert scale: definitely yes; probably yes; probably no; definitely no.. See attached protocol.

SECONDARY OUTCOMES:
Understanding | Assessed during 15-minute survey.
  Multiple choice questions assessing participants understanding of the information in the patient leaflet (e.g., what is Fotivda used for?)
  Each question includes several response options, with 1 correct answer per item. See attached protocol.
Perceived magnitude of benefits and harms | Assessed during 15-minute survey
  Multiple choice questions assessing participants perceived magnitude of the drug's benefits and harms (e.g., Overall, how large are the benefits of Fotivda?)
  Likert scales vary depending on the question. See attached protocol.
Satisfaction with information in the patient leaflet | Assessed during 15-minute survey.
  Multiple choice questions assessing participants' satisfaction with information included in the patient leaflet (e.g., ease of finding and understanding information).
  Likert scales vary depending on the question. See attached protocol.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-07-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT07061197/Prot_SAP_ICF_000.pdf